CLINICAL TRIAL: NCT02714712
Title: Influence of Scavenger Receptor Class B Type I (SR-BI) Gene Polymorphisms on Antiviral Treatment Response, and Metabolism in Chronic Hepatitis C Patients
Brief Title: SR-BI and Antiviral Treatment Response in HCV
Status: Completed | Type: Observational
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Ching-Sheng Hsu, Attending physician, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Other Study IDs: 03-XD53-105
Record Dates: First submitted 2016-03-09; First posted 2016-03-21 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — All enrolled subjects were genotyped for the SNPs of the SCARB1 gene and IL28B gene. All their blood specimens were collected into EDTA tubes. Human genomic DNA was extracted by standard protocols with blood RBC lysis, cell lysis, DNA binding, wash and elution. Extracted DNA normalized to 50 ng/µl was obtained. DNA quality was assessed by calculating the absorbance ratio OD260 nm/280 nm using NanoDrop model ND-1000 (Thermo Scientific, Wilmington, DE, USA). The SNP was genotyped by using the ABI TaqMan allelic discrimination kit and the ABI7900HT Sequence Detection System (Applied Biosystems, Foster City, CA, USA)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HCV group (Peginterferon alfa-2a): A total of 156 chronic HCV genotype 1 or 2 patients who received Peginterferon alfa-2a (Peg-IFN alfa-2a) plus ribavirin therapy were consecutively enrolled from the gastroenterological clinics.
  Interventions: Drug: Peginterferon alfa-2a
- Control Group: There were 153 healthy controls negative for anti-HCV enrolled simultaneously from the database of Health Management Center.

INTERVENTIONS:
Drug: Peginterferon alfa-2a — Peginterferon alfa-2a 180μg plus daily oral weight-based ribavirin (1,000 mg for body weight 75 kg or less, 1,200 mg for body weight greater than 75 kg) for 24 or 48 weeks
  Other Names: Pegsys
  Groups: HCV group (Peginterferon alfa-2a)

SUMMARY:
The scavenger receptor type B class I (SR-BI) is a receptor for high-density lipoproteins (HDL) and one of entry factors for hepatitis C virus (HCV). The investigators aimed to examine the association of single nucleotide polymorphisms (SNPs) of the SCARB1 gene, which encodes SR-BI, with virologic responses to pegylated interferon-based treatment in Asian chronic hepatitis C (CHC) patients.

DETAILED DESCRIPTION:
1. Purpose of study: To examine the impacts of single nucleotide polymorphisms (SNPs) relevant to SR-BI on CHC patients.
2. Study Design To enroll 400 CHC patients during a 3-year period
3. Specify objectives of study when collecting extra specimen from participants Collect blood samples for genomic DNA to examine the SR-BI gene polymorphisms.
4. Expected Endpoints of Treatment Sustained virologic response (SVR) means undetectable serum HCV RNA levels 24 weeks after completion of antiviral therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Naive to IFN treatment and other experimental antiviral or immunosuppressive therapy before enrollment.
2. Serum alanine aminotransferase levels, at least, twice the upper limit of normal on two occasions within the previous 6 months.

Exclusion Criteria:

1. Positive for hepatitis B surface antigen
2. Positive for human immunodeficiency virus antibody
3. Had a known history or evidence of autoimmune liver disease, inheritable disorders, renal insufficiency, malignancy
4. Had a history of daily alcohol consumption greater than 20 gram or active drug abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCV genotype 1 or 2 patients who received pegylated interferon alfa-2a (Peg-IFN alfa-2a) plus ribavirin therapy were consecutively enrolled from the gastroenterological clinics
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Serum HCV RNA levels | at 24 weeks after the end of treatment
  sustained virologic response

SECONDARY OUTCOMES:
serum fasting blood glucose levels | at 24 weeks after the end of treatment

IPD SHARING:
Plan to Share IPD: Yes
Share data when requested

REFERENCES:
- [Derived] Hsu CS, Hsu SJ, Liu WL, Chen DS, Kao JH. Association of SCARB1 Gene Polymorphisms with Virological Response in Chronic Hepatitis C Patients Receiving Pegylated Interferon plus Ribavirin Therapy. Sci Rep. 2016 Aug 26;6:32303. doi: 10.1038/srep32303. PMID 27561198